CLINICAL TRIAL: NCT06088628
Title: Study of Micro-expressions in Patients With Prolonged Disorders of Consciousness
Brief Title: Micro-expressions in Patients With Prolonged Disorders of Consciousness
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Hangzhou Mingzhou Brain Rehabilitation Hospital (Unknown); Zhejiang Provincial People's Hospital (Other); Zhejiang Provincial Armed Police Corps Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: Micro-expression
Record Dates: First submitted 2023-08-29; First posted 2023-10-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Consciousness Disorders
Keywords: disorders of consciousness; consciousness disorders; microexpressions; emotional stimuli; consciousness
MeSH Terms: conditions — Consciousness Disorders | interventions — Electroencephalography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DoC patients: Patients with disorders of consciousness.
  Interventions: Diagnostic Test: Facial expression; Electroencephalogram; MRI
- Healthy controls: Healthy participants matched by gender and age.
  Interventions: Diagnostic Test: Facial expression; Electroencephalogram; MRI

INTERVENTIONS:
Diagnostic Test: Facial expression; Electroencephalogram; MRI — Recording facial expressions of participants, EEG recordings, and MRI scans.

SUMMARY:
The goal of this observational study is to learn about the microexpressions in patients with prolonged disorders of consciousness. The main questions it aims to answer are:

* Inducing micro-expression changes in patients with prolonged disorders of consciousness through various emotional stimuli, and further to achieve precise classification of their levels of consciousness.
* Detecting micro-expressions in patients with prolonged disorders of consciousness to assist clinical diagnosis of levels of consciousness, e.g., complement the disgnosis of clinical scales such as CRS-r scale.
* By monitoring micro-expression changes in patients with prolonged disorders of consciousness, researchers can explore their residual brain function, thereby advancing research into relevant neural mechanisms.

Participants will be subjected to consciousness assessment by CRS-r scale, and their micro-expression changes in response to various emotional stimuli will be captured, along with the collection of EEG and MRI data. Follow-up evaluations will be conducted using the CRS-R scale and GOS scale, with a follow-up period of 6 months.

DETAILED DESCRIPTION:
In accordance with the inclusion and exclusion criteria, a total of about 200 participants will be recruited, including about 150 confirmed cases of prolonged disorders of consciousness and 50 healthy control subjects (HCs). Utilizing the random split algorithm from the machine learning library sklearn, the dataset will be randomly divided into a training set (70%) and a testing set (30%). General information about the participants such as age, gender, time and location of injury, as well as medical history, family history, medication history, and surgical history will be collected.

Participants will undergo dual-person, multiple assessments using the CRS-R scale to evaluate auditory, visual, motor, speech responsiveness, communication, and arousal levels. Micro-expression changes in response to various emotional stimuli will be collected, along with EEG and MRI data.

Follow-up evaluations will be conducted on all enrolled patients using the CRS-R scale and the GOS scale, with a follow-up period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with consciousness disorders for more than 28 days following severe brain injury, assessed by the CRS-R scale to meet the criteria for VS or MCS;
2. Aged between 18 and 80 years;
3. Stable vital signs;
4. Voluntary participation of family members with signed informed consent;
5. Good cooperation, minimal facial and spontaneous activities, no use of antiepileptic or sedative drugs.

Exclusion Criteria:

1. Locked-in syndrome;
2. Contraindications for EEG examination;
3. Contraindications for MRI scanning, such as the presence of internal metallic implants;
4. Diseases and factors that may affect brain function assessment, such as metabolic disorders, poisoning, shock, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from both general hospitals and rehabilitation hospitals.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
GOSE score | six month
  GOS-E is an extended version of the Glasgow Outcome Scale (GOS), which was developed to provide a more detailed assessment of patient functionality and quality of life after experiencing such an injury. It has eight categories: Dead, Vegetative State, Lower Severe Disability, Upper Severe Disability, Lower Moderate Disability, Upper Moderate Disability, Lower Good Recovery, and Upper Good Recovery
CRS-r score | six month
  CRS-R a standardized neurobehavioral assessment measure designed for use in patients with disorders of consciousness. The scale is intended to be used to establish diagnosis, monitor behavioral recovery, predict outcome, and assess treatment effectiveness. The CRS-R consists of 6 subscales designed to assess auditory function, receptive and expressive language, visuoperception, communication ability, motor functions, and arousal level.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Doctor, Principal Investigator — Zhejiang University
Locations (1):
- First Affiliated Hospital,Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided